CLINICAL TRIAL: NCT04431037
Title: EARLY ORAL FEEDING VS TRADITIONAL POST-OPERATIVE CARE IN PATIENTS UNDERGOING EMERGENCY ABDOMINAL SURGERY FOR PERFORATED DUODENAL ULCER(Emergency Abdominal Surgeries)
Brief Title: Early Oral Feeding vs Traditional Post-operative Care In Emergency Abdominal Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: College of Physicians and Surgeons Pakistan (Other)
Responsible Party: Principal Investigator, Ayesha Masood, Postgraduate trainee, General Surgery, College of Physicians and Surgeons Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: pdu
Record Dates: First submitted 2020-06-03; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Perforated Duodenal Ulcer
Keywords: Perforated duodenal ulcer; Enhanced Recovery After Surgery (ERAS) protocol; Randomized controlled trial; Duodenal repair site leak; Length of hospital stay; Visual analog score; Post-operative ileus

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial was conducted in Surgical Unit 1 BBH from August 2018 to December 2019 with a total sample size of 36 patients with the diagnosis of perforated duodenal ulcer. Patients were randomly divided in two groups. Group A consisted of early oral feeding group and group B consisted of traditional postoperative care group. Outcome results studied were the length of hospital stay, duodenal repair site leak, severity of pain (VAS score) and duration of post-operative ileus. Results were analysed on SPSS version 20 and chi-square and independent t-test were applied.
Who Masked: Participant, Investigator
Masking Description: Patients admitted in the emergency department were randomly assigned into treatment group or control group in postoperative period.Neither the researcher nor the patient were aware of the patient allocation.Patients were management by the oncall surgical team irrespective of the researcher.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early oral feeding group(A) (Experimental): Patients admitted in the HDU postoperatively.NG tube and foley's catheter removed within 12 hours and patients allowed oral sips on day 1 with gradual shift to liquid diet after 12 hrs and semisolid food started after 24 hours later.Patients were given i/v antibiotics,painkillers and i/v PPIs and shifted to oral pain killers on 2nd POD.
  Interventions: Dietary Supplement: Early oral feeding/Enhanced recovery after surgery protocols
- Traditional postoperative care group(B) (No Intervention): Patients in this group were managed traditionally

INTERVENTIONS:
Dietary Supplement: Early oral feeding/Enhanced recovery after surgery protocols — Early oral feeding refers to NG tube and foley's catheter removed within 12 hours and patients allowed oral sips on day 1 with gradual shift to liquid diet after 12 hrs and semisolid food started after 24 hours later.Patients were given i/v antibiotics,painkillers and i/v PPIs and shifted to oral pain killers on 2nd POD.
  Arms: Early oral feeding group(A)

SUMMARY:
ABSTRACT BACKGROUND: Enhanced recovery after surgery (ERAS) protocols have been widely studied in elective abdominal surgeries and have shown better outcomes. However the utility of these protocols in emergency abdominal surgeries has not been widely investigated.

OBJECTIVE: To study the outcomes of application of ERAS protocols in patients undergoing perforated duodenal ulcers repairs in emergency abdominal surgeries.

METHODS: This randomized controlled trial was conducted in Surgical Unit 1 BBH from August 2018 to December 2019 with a total sample size of 36 patients with the diagnosis of perforated duodenal ulcer. Patients were randomly divided in two groups. Group A consisted of early oral feeding group and group B consisted of traditional postoperative care group. Outcome results studied were the length of hospital stay, duodenal repair site leak, severity of pain (VAS score) and duration of post-operative ileus. Results were analysed on SPSS version 20 and chi-square and independent t-test were applied.

KEY WORDS: Perforated duodenal ulcer, ERAS protocol, randomized controlled trial, duodenal repair site leak, length of hospital stay, VAS score, post-operative ileus

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 15 years with acute abdominal symptoms admitted in ER department, suspected as perforated duodenal ulcer and operated within 24 hours of admission by emergency department surgeon.

Exclusion Criteria:

* Patients presenting with the following criteria were excluded:
* Refusal to join the study
* Peptic ulcers with both bleeding and perforation.
* Spontaneously sealed off perforations.
* Malignant ulcers
* Concurrent extra-abdominal surgery
* Oral incapacity i.e endotracheal intubation
* Reoperation within a month
* ASA grade III/IV
* Alternative per operative diagnosis.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | upto 10 Days
  Length of hospital stay is defined as duration of single episode of hospitalization. Inpatient days are calculated by subtracting day of admission from day of discharge
DAYS OF RETURN OF BOWEL FUNCTION. | Upto 24 hours
  It is defined as time to passage of flatus or stools after abdominal surgery.
Pain score by Visual Analog Scale | upto 36 hours
  Pain is defined as "an unpleasant sensory and emotional experience that is associated with actual or potential tissue damage or described in such terms" according to International Association for the Study of Pain,measured by Visual Analog Scale(VAS).

SECONDARY OUTCOMES:
Bleeding peptic ulcer | intraoperative period
  Frequency of bleeding peptic ulcer
Mortality rate | immediate postoperative period
  Estimation of mortality rate associated with perforated duodenal ulcer

OTHER OUTCOMES:
Gender distribution | Perioperative period
  To assess the frequency of perforated duodenal ulcer according to gender

CONTACTS AND LOCATIONS:
Locations (1):
- Surgical Unit I,Benazir Bhutto Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on request.Only that described in the text of full article.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-08-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT04431037/Prot_SAP_ICF_000.pdf